CLINICAL TRIAL: NCT03545971
Title: A Phase I, Open-Label Study to Investigate the Tolerability and Safety of IBI310 Alone or in Combination With Sintilimab in the Treatment of Patients With Advanced Solid Tumors.
Brief Title: A Study of IBI310 for the Treatment of Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310A101
Record Dates: First submitted 2018-05-10; First posted 2018-06-06 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — CTLA-4 Antigen; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Ia Cohort A (Experimental): Low-dose group:Participants will receive IBI310 0.3mg/kg intravenous every 3 weeks,after 4 cycle, if the patient benefits it will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: IBI310
- Ia Cohort B (Experimental): Middle-dose group:Participants will receive IBI310 1.0mg/kg intravenous every 3 weeks,after 4 cycle, if the patient benefits it will be continued until disease progression or unacceptable toxicity
  Interventions: Drug: IBI310
- Ia Cohort C (Experimental): Middle-dose group:Participants will receive IBI310 2.0mg/kg intravenous every 3 weeks,after 4 cycle, if the patient benefits it will be continued until disease progression or unacceptable toxicity
  Interventions: Drug: IBI310
- Ia Cohort D (Experimental): High-dose group:Participants will receive IBI310 3.0mg/kg intravenous every 3 weeks,after 4 cycle, if the patient benefits it will be continued until disease progression or unacceptable toxicity
  Interventions: Drug: IBI310
- Ib Cohort A (Experimental): 3 subjects, low-dose group:Participants will receive IBI310 1.0mg/kg in Combination with Sintilimab 200mg intravenous every 3 weeks. After 4 cycles, Sintilimab alone 200mg intravenous every 3 weeks, until disease progression, lost follow-up visit, death , unacceptable toxicity, withdrawn of ICF, another other reason for end of treatment. Maximum treatment duration is 2 years.
  Interventions: Drug: IBI310; Drug: Sintilimab
- Ib Cohort A2 (Experimental): low-dose group:Participants will receive IBI310 1.0mg/kg in Combination with Sintilimab 200mg intravenous every 3 weeks. After 4 cycles, Sintilimab alone 200mg intravenous every 3 weeks, until disease progression, lost follow-up visit, death , unacceptable toxicity, withdrawn of ICF, another other reason for end of treatment. Maximum treatment duration is 2 years.
  Interventions: Drug: IBI310; Drug: Sintilimab
- Ib Cohort B (Experimental): 3 subjects, low-dose group:Participants will receive IBI310 2.0mg/kg in Combination with Sintilimab 200mg intravenous every 3 weeks. After 4 cycles, Sintilimab alone 200mg intravenous every 3 weeks, until disease progression, lost follow-up visit, death , unacceptable toxicity, withdrawn of ICF, another other reason for end of treatment. Maximum treatment duration is 2 years.
  Interventions: Drug: IBI310; Drug: Sintilimab
- Ib Cohort B2 (Experimental): low-dose group:Participants will receive IBI310 2.0mg/kg in Combination with Sintilimab 200mg intravenous every 3 weeks. After 4 cycles, Sintilimab alone 200mg intravenous every 3 weeks, until disease progression, lost follow-up visit, death , unacceptable toxicity, withdrawn of ICF, another other reason for end of treatment. Maximum treatment duration is 2 years.
  Interventions: Drug: IBI310; Drug: Sintilimab

INTERVENTIONS:
Drug: IBI310 — IBI310 is anti CTLA-4 antibody
  Other Names: CTLA-4
Drug: Sintilimab — PD-1 monoclonal antibody
  Arms: Ib Cohort A; Ib Cohort A2; Ib Cohort B; Ib Cohort B2

SUMMARY:
This is an open-label, dose escalation, Phase I study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity and efficacy of single agent of IBI310, and in combination of sintilimab, in patients with advanced solid tumors(Ia) and advanced melanoma(Ib).

DETAILED DESCRIPTION:
Phase Ia study will adopt the classical 3+3 dose escalation design. The starting dose is 0.3 mg/kg, followed by 3 dose cohorts (1mg/kg, 2mg/kg and 3mg/kg). Duration of dose limiting toxicity (DLT) observation period is 21 days. IBI310 treatment q3w, up to 3 cycles, will be provided to patients who complete DLT observation period.

Efficacy will primarily be evaluated by RECIST v1.1. Patient safety will be monitored throughout the study. Pharmacokinetic/pharmacodynamics and immunogenicity will be assessed throughout the study.

Phase Ib study will evaluate the tolerability and safety of IBI310 combined with Sintilimab in patients with advanced melanoma. Phase Ib of the study will begin after DLT observation is completed in certain dose cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with locally advanced, recurrent or metastatic solid tumors who failed standard treatment(applicable to the Ia period).
2. Patients with advanced, recurrent or metastatic melanoma confirmed by cytology or histology (applicable to the Ib period).
3. Signed written informed consent form and willing and able to comply with scheduled visits and other requirements of the study.
4. ≥18，and ≤70 years.
5. Life expectancy of at least 12 weeks.
6. At least 1 measurable lesion per RECIST v1.1(long axis>15mm or short axis>10mm)
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1.
8. Patients of reproductive potential must be willing to use adequate contraception during the course of the study and through 6 months after the last dose of study medication.
9. Adequate organ and bone marrow function.

Key Exclusion Criteria:

1. Prior exposure to any anti-CTLA-4, anti-PD-1 or anti-PD-L1/L2 antibody.
2. Received any investigational agent within 4 weeks of the first dose of study medication.
3. Received last dose of anti-tumor therapy (chemotherapy, endocrine therapy, targeted therapy, tumor immunotherapy or arterial embolization) within 4 weeks of the first dose of study medication.
4. Received treatment with corticosteroids (>10mg daily prednisone equivalent) or other immunosuppressive medications within 4 weeks before the first dose of study medication. Nasal spray, inhalation, or other ways of topical corticosteroids or physiological doses of systemic corticosteroids are not included.
5. Received a live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during study period.
6. Active, known or suspected autoimmune disease or has a history of the disease within the last 2 years (Patients with vitiligo, psoriasis, alopecia or Grave's disease, hypothyroidism requiring hormone replacement, or type I diabetes mellitus only requiring insulin replacement, but not required systemic treatment in the last 2 years, are permitted to enroll)
7. Known primary immunodeficiency
8. Active tuberculosis
9. Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation
10. Known allergy or hypersensitivity to any other monoclonal antibodies or IBI310 and/or any components used in their preparation.
11. Known acute or chronic active hepatitis B (HBV DNA positive and HBV DNA copies ≥1×103/ml or ≥200IU/ml) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection. Patients with HCV antibody positive but HCV RNA negative are permitted to enroll.
12. Patients with a history of interstitial lung disease
13. Uncontrolled third space effusion, eg. ascites or pleural effusion cannot be drained or controlled.
14. Women who are pregnant or nursing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
AEs | up to 24 months after randomization
  Number of patients with treatment-related adverse events (AEs)

SECONDARY OUTCOMES:
Pharmacokinetics：Cmax | up to 24 months after randomization
  Maximum concentration(Cmax) of the drug after administration
pharmacodynamics:lipid parameters | up to 24 months after randomization
  Change from baseline in lipid parameters
ADA | up to 24 months after randomization
  Number of participants with anti-drug antibodies or neutralizing antibodies
Pharmacokinetics：AUC | up to 24 months after randomization
  The area under the curve (AUC) of serum concentration of the drug after the administration

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China